CLINICAL TRIAL: NCT00619528
Title: HLA-Identical Sibling Renal Transplant Tolerance With Donor Hematopoietic Stem Cells and Campath-1H
Brief Title: HLA-Identical Sibling Renal Transplant Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joseph Leventhal, Professor, Department of Surgery, Division of Organ Transplantation, Feinberg School of Medicine; Director, Kidney Pancreas Program, Comprehensive Transplant Center, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2R01DK025243-25A2 (NIH); R01DK025243 (NIH)
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Immunosuppression; Kidney Transplantation; Graft Rejection
Keywords: Transplants; Kidney Transplantation; Immunosuppression; HLA Antigens; Stem Cells; Bone Marrow
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): No separate arms: All Enrolled Receive Same Treatment
  Interventions: Biological: Infusion of Donor Hematopoietic Stem Cells and Campath-1H

INTERVENTIONS:
Biological: Infusion of Donor Hematopoietic Stem Cells and Campath-1H — Intervention: a four-dose (peri-operative and 3, 6, and 9-month boost) DHSC infusion protocol using two-dose Campath-1H induction combined with transient (conditioning) Tacrolimus/Sirolimus and MMF therapy will result in a high degree of macro-chimerism (>10%), and a robust prolonged donor-specific (post-thymic) immunoregulatory condition that will allow renal transplant survival in the absence of permanent immunosuppression.

SUMMARY:
The purpose of this study is to attempt to eliminate the necessity of immunosuppressive therapy for HLA-identical sibling Kidney Transplants, examine cellular chimerism of donor hematopoietic stem cell (DHSC) lineages for pairs to demonstrate immunologic unresponsiveness, and to investigate the safety and efficacy of the treatment regimen including withdrawal of immunosuppression after one year post-transplant for those recipients having received DHSC infusions.

DETAILED DESCRIPTION:
Primary Study Objectives:

1. To remove all immunosuppressive therapy from recipients of HLA-identical sibling renal transplants within 24 months of transplantation.
2. To detect and follow cellular (macro) chimerism of donor hematopoietic stem cell (DHSC) lineages and the generation of T-regulatory cells using specialized immunomonitoring assays for these donor/recipient pairs to demonstrate specific immunologic unresponsiveness.
3. To investigate the safety and efficacy of a treatment regimen consisting of induction therapy with Campath-1H and steroid-free low dose maintenance immunosuppression, consisting of mycophenolate mofetil (MMF) and tacrolimus converted to sirolimus. This is to be followed by complete withdrawal of immunosuppression beginning at one year, at a minimum, post transplant, in recipients who have also been given four infusions of purified donor hematopoietic Cluster of Differentiation (CD)34+ stem cells (DHSC).

ELIGIBILITY:
Inclusion Criteria:

* Patient fully informed, signed dated Institutional Review Board (IRB)-approved informed consent form obtained directly by the P.I., Co-P.I., or Res. Nurse, and willing to follow study procedures for the duration of study (3 yrs).
* Recipient: a hematocrit of ≥ 33%, and a hemoglobin of ≥ 11.0 g/dL.
* Weight > 40 kg.
* Primary renal allograft: living related (HLA-identical donor-recipient sibling pairs)
* Negative B-cell and T-cell cytotoxic cross-match, and a low (≤ 10%) Panel Reactive Antibody (PRA) using cytotoxicity.
* Women of childbearing potential: negative qualitative serum pregnancy test.
* Patients studied equivalently as available for transplant using criteria, w/out regard to gender, race, or ethnicity.
* Normal echocardiogram w/ ejection fraction >50%.
* Male participants w/ reproductive potential agree to use approved methods of birth control during treatment w/ Campath-1H and for minimum of 6 months following last dose. Female participants of childbearing potential agree to use approved methods of birth control for duration of participation in study.
* Patient agrees to follow-up every 2 months after year 3, up to 10 years.

Exclusion Criteria:

* Patient previously received/receiving transplant other than kidney.
* Patient receiving ABO (blood type) incompatible donor kidney.
* Recipient/donor is ELISA positive for human immunodeficiency virus (HIV), antibody positive for hep. C, or surface antigen positive for hep. B.
* Patient has current malignancy or history of malignancy (within past 5 years), except non-metastatic basal or squa¬mous cell carcinoma of the skin, or carcinoma in situ of the cervix that has been treated successfully.
* Patients w/ significant liver disease, defined as having during past 28 days continuously elevated aspartate aminotransferase (AST (SGOT)) and/or Alanine Aminotransferase (ALT (SGPT)) levels greater than 3 times the upper value of the normal range at this center.
* Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer or other unstable medical condition that could interfere w/ study objectives.
* Patient currently receiving investigational drug or received an investigational drug within 30 days pre-transplant.
* Patient currently receiving immunosuppressive agent.
* In investigator's judgment, anticipated that patient unable to take medications orally or via nasogastric tube by morning of second day (i.e., skin closure).
* Concurrent use of warfarin, fluvastatin, astemizole, pimozide, cisapride, terfenadine, or ketoconazole.
* Patient hypersensitivity to tacrolimus, Campath-1H, Thymoglobulin, daclizumab (Zenapax®), sirolimus, MMF or corticosteroids.
* Patient pregnant or lactating.
* Patients w/ screening/baseline total white blood cell count <4000/mm3; platelet count <100,000/mm3; fasting triglycerides >400 mg/dl (>4.6 mmol/L); fasting total cholesterol >300 mg/dl (>7.8 mmol/L); fasting HDL-cholesterol <30 mg/dl; fasting LDL-cholesterol >200 mg/dl.
* Patient unlikely to comply w/ visits.
* Patient w/ any form of substance abuse, psychiatric disorder or condition that, in investigator's opinion, may invalidate communication.
* Expected that tacrolimus cannot be instituted for over 5 days post-operatively.
* Patients w/ cytotoxic PRA value >10% any time pre-enrollment.
* Patients w/ Graves disease, unless previously treated w/ radioiodine ablative therapy.
* History of idiopathic thrombocytopenic purpura (ITP) or thrombotic thrombocytopenic purpura (TTP)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2023-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leventhal, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Derived] Leventhal JR, Mathew JM, Salomon DR, Kurian SM, Friedewald JJ, Gallon L, Konieczna I, Tambur AR, Charette J, Levitsky J, Jie C, Kanwar YS, Abecassis MM, Miller J. Nonchimeric HLA-Identical Renal Transplant Tolerance: Regulatory Immunophenotypic/Genomic Biomarkers. Am J Transplant. 2016 Jan;16(1):221-34. doi: 10.1111/ajt.13416. Epub 2015 Jul 30. PMID 26227106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment 2008-2012. Subjects were recruited at the Northwestern University Medical Center, in the comprehensive Transplant Center.
  Enrollment has been completed since 2012
Pre-assignment Details: 1 subject did not did not receive the DHSC infusions due to the immediate pre-operative cross-match again the donor that was unexpectedly found to be positive
Groups:
- Experimental: Recipients of Infusion of Donor Hemopoietic Steam Cells (n=20)
- Donor: Donor of HLA identical donor-recipient sibling pairs
- Healthy Controls: Healthy Controls do not have the disease or problem being studied.
- Parents of Recipients/Donors: Parent(s) to donor/recipient children
Period: Overall Study
Arm/Group | Experimental | Donor | Healthy Controls | Parents of Recipients/Donors
Started | 20 | 20 | 19 | 29
Completed | 19 | 0 | 0 | 0
Not Completed | 1 | 20 | 19 | 29

BASELINE CHARACTERISTICS:
Population: Recipient, Donor, Healthy Controls & Parents of recipients/donors
Groups:
- Recipients: Recipient of kidney transplant
- Donor: Donating kidney to sibling
- Healthy Controls: The control subjects (not having the disease or problem being studied) either have a one time bone marrow aspiration (taking bone marrow out of one or both hip bones) and/or having blood taken for the study.
- Parents of Recipients/Donors: The subjects in this group are the parents of donors and recipients of kidney transplant
- Total: Total of all reporting groups
Arm/Group | Recipients | Donor | Healthy Controls | Parents of Recipients/Donors | Total
Number analyzed (Participants) | 20 | 20 | 19 | 29 | 88
Age, Continuous [Mean (Full Range); unit: years] | 39.625 [20 to 54] | 39.241 [19 to 53] | 36.034 [19 to 74] | 53.379 [42 to 74] | 36.034 [19 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 9 | 17 | 41
  Male | 16 | 9 | 10 | 12 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 6 | 11
  Not Hispanic or Latino | 17 | 17 | 16 | 23 | 73
  Unknown or Not Reported | 0 | 1 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 3 | 3 | 3 | 3 | 12
  White | 14 | 13 | 8 | 20 | 55
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 3 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Ability to Withdraw Immunosuppression as Above 24 Months Post-transplant
Description: The ability to withdraw immunosuppression as above 24 months post-transplant with follow-up to 10 years.
Time Frame: 24 months post-transplant with follow-up to 10 years
Measure: Count of Participants; unit: Participants
Groups:
- Kidney Transplant Recipients Who Received Infusion of Donor Hematopoietic Stem Cells and Campath-1H: No separate arms: All Enrolled Receive Same Treatment
  Infusion of Donor Hematopoietic Stem Cells and Campath-1H: Intervention: a four-dose (peri-operative and 3, 6, and 9-month boost) DHSC infusion protocol using two-dose Campath-1H induction combined with transient (conditioning) Tacrolimus/Sirolimus and MMF therapy will result in a high degree of macro-chimerism (>10%), and a robust prolonged donor-specific (post-thymic) immunoregulatory condition that will allow renal transplant survival in the absence of permanent immunosuppression.
Arm/Group | Kidney Transplant Recipients Who Received Infusion of Donor Hematopoietic Stem Cells and Campath-1H
Number analyzed (Participants) | 19
Participants | 6

2. Primary Outcome: Patient and Graft Survival
Description: Patient and graft survival measured at the one-year timepoint post-transplant.
Time Frame: One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Kidney Transplant Recipients Who Received Infusion of Donor Hematopoietic Stem Cells and Campath-1H
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Over 10 year after receiving consenting to the study
Groups:
- Recipient of Transplant: Recipient with Infusion of Donor Hematopoietic Stem Cells and Campath-1H:
- Healthy Controls: Control subjects (not having the disease or problem being studied) either have at one time bone marrow aspiration (taking bone marrow out of one or both hip bones) and/or having blood taken for the study
- Parents of Recipients/Donors: The subjects in this group are the parents of the donor and recipient of kidney transplant
Arm/Group | Recipient of Transplant | Donor | Healthy Controls | Parents of Recipients/Donors
All-Cause Mortality (participants affected / at risk) | 4/20 | 0/20 | 0/19 | 0/29
Serious Adverse Events (participants affected / at risk) | 8/20 | 0/20 | 0/19 | 0/29
Other Adverse Events (participants affected / at risk) | 4/20 | 0/20 | 0/19 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipient of Transplant (N=20) | Donor (N=20) | Healthy Controls (N=19) | Parents of Recipients/Donors (N=29)
Pancreatic Neuroendocrine Tumor (Endocrine disorders) | 1 (1) | NA | NA | NA — Pancreatic Neuroendocrine Tumor (Determined to be unrelated to study product)
Prostrate Cancer (Renal and urinary disorders) | 1 (1) | NA | NA | NA — Prostrate Cancer ((Determined to be unrelated to study product)
Hospitalizations (General disorders) | 4 (4) | NA | NA | NA — (Determined to be unrelated to study product)
Acute Tubular Necrosis (Renal and urinary disorders) | 1 (1) | NA | NA | NA
Severe Cellular Rejection (Renal and urinary disorders) | 1 (1) | NA | NA | NA
Heart Failure (Cardiac disorders) | 1 (1) | NA | NA | NA — (Determined to be unrelated to study product)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipient of Transplant (N=20) | Donor (N=20) | Healthy Controls (N=19) | Parents of Recipients/Donors (N=29)
UTI (Renal and urinary disorders) | 1 (1) | NA | NA | NA — Determined not be be related to study drug
Allergic Reaction following second dose of Altuzemab (Product Issues) | 3 (3) | NA | NA | NA

LIMITATIONS AND CAVEATS:
20 Donor Recipient Pairs were enrolled (n=40)

In addition, 19 controls and 29 parents were also enrolled.

This study was concluded earlier than anticipated due to changes in funding support, which impacted the ability to meet all originally stated enrollment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT00619528/Prot_SAP_000.pdf